CLINICAL TRIAL: NCT01906606
Title: Effectiveness of Parenting Programs on Child Development and Maternal Well-being in Rural Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Mbarara University of Science and Technology (Other)
Responsible Party: Principal Investigator, Frances Aboud, Professor, McGill University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: REB#231-1112
Record Dates: First submitted 2013-07-03; First posted 2013-07-24 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Child Development; Depression
Keywords: child nutritional status; child development; maternal depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parenting Program (Experimental): 12 session community-based parenting program
  Interventions: Behavioral: Parenting Program
- Control Group (No Intervention): received visual aids on nutrition

INTERVENTIONS:
Behavioral: Parenting Program — A manualized, community-based 12 session group parenting program, facilitated by a locally recruited volunteer
  Arms: Parenting Program

SUMMARY:
The purpose of the current study involves the development, implementation and evaluation of a parenting program to target maternal well-being and child health, growth and development in Lira, Uganda. The current study aims to address maternal care within a parenting program as well as parenting practices emphasizing nutrition, hygiene, and psychosocial stimulation through peer-support, practice and problem-solving. Outcomes include child health, growth and development, maternal mental health, mother-child interactions, and maternal-spousal relations.

We hypothesize that:

1. Children of parents who attend the parenting program will have better health, height and cognitive/language development at post-test, than children whose parents did not have the opportunity to attend parenting sessions.
2. Parents who attend the parenting program will have more knowledge about child development and provide more home stimulation, dietary diversity and preventive health practices than parents who do not have the opportunity to attend parenting sessions.
3. Mothers who attend the parenting program will have improved well-being compared to mothers who do not have the opportunity to attend parenting sessions.

ELIGIBILITY:
Inclusion Criteria:

* mothers of children ages 12-24 months

Exclusion Criteria:

* disabled children

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Bayley III Language scale | Baseline and 11 months
  receptive and expressive language subtests

SECONDARY OUTCOMES:
Change from baseline in CES-D | Baseline and 11 months
  maternal depressive symptoms (CES-D) and perceived positive and negative support

OTHER OUTCOMES:
Change from Baseline in child length-for-age | Baseline and 11 months
  length for age

CONTACTS AND LOCATIONS:
Overall Officials: Frances Aboud, PhD, Principal Investigator — McGill University
Locations (1):
- Lira Program Unit, Plan Uganda, Lira, Uganda

REFERENCES:
- [Derived] Singla DR, Kumbakumba E, Aboud FE. Effects of a parenting intervention to address maternal psychological wellbeing and child development and growth in rural Uganda: a community-based, cluster randomised trial. Lancet Glob Health. 2015 Aug;3(8):e458-e469. doi: 10.1016/S2214-109X(15)00099-6. Epub 2015 Jul 2. PMID 26144389